CLINICAL TRIAL: NCT06364579
Title: Patient Reported Outcomes (PROs) in Anal Cancer Patient Treated by Intensity Modulated Radiotherapy (IMRT).
Acronym: PROACT
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Manfrida Stefania, Radiation oncologist, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 6533
Record Dates: First submitted 2024-03-28; First posted 2024-04-15 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Anal Cancer Patients
Keywords: PROs; QOL; EORTC; anal cancer; radiotherapy; radiation therapy; follow up
MeSH Terms: conditions — Anus Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Radiochemotherapy is the standard treatment for neoplasms of the anal canal with excellent rates of local control and preservation of the anal sphincter. However, patients may experience a deterioration of quality of life related to sequelae of the treatment particularly at intestinal, anal sphincter and sexual level. Few studies to date have documented patient-reported outcomes (PROs) in this area. The aim of this observational study is to verify the quality of life (QOL) of the patients by means of self-completed questionnaires.

DETAILED DESCRIPTION:
In recent times, the focus on collecting patient-reported outcomes (PROs) has increased in healthcare. The Food and Drug Administration defines PROs as a -measurement of any aspect of a health status of the patient that comes directly from the patient-. These includes disease symptoms, functional aspects and quality of life (QOL). The collection of PROs, combined with physician-assessed toxicity, is constantly being incorporated into clinical practice and studies to provide a more holistic picture of the impact of treatment on patients and prove useful for planning future interventions. Although the use of PROs has now become the standard for measuring quality of life of patients there are still few studies on the self-reported long-term QOL of anal cancer patients and on disease or therapy related symptoms that affect QOL. Therefore, the EORTC (European Organisation for Research and Treatment of Cancer) has recently developed the specific Quality of Life Questionnaire for anal cancer (QLQ-AN27) module to explore typical symptoms of anal cancer and its therapy. In this study, the QLQ-AN27 questionnaire will be administered together with the EORTC Quality of Life 30 (QLQ 30) in patients with anal cancer who have undergone radio-chemotherapy. The questionnaire may be administered before treatment, after treatment and during follow-ups until completion of the fifth year. This is an observational study both retrospective and prospective.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) 0-3
* minimum 18 years old
* squamous cell carcinoma of the anal canal
* low burden of metastatic disease at diagnosis
* indication for radiochemotherapy treatment
* informed consent

Exclusion Criteria:

* age under 18 years
* Eastern Cooperative Oncology Group (ECOG) higher than 3
* metastatic disease at diagnosis not amenable to radiochemotherapy treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with anal cancer treated with radiochemotherapy at the Fondazione Policlinico Gemelli from 2010 to the present.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-03-28 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2031-01-31 (Estimated)

PRIMARY OUTCOMES:
QOL analysis | 60 months from the last enrolled patient (january 2026)
  Analysis of quality of life (QOL) by administration of PRO questionnaires to patients with cancer of the anus treated with IMRT radiochemotherapy.

SECONDARY OUTCOMES:
Overall survival (OS) | time 0, end of treatment, 6 month post treatment, 1 year follow-up, 2 years follow-up, 3 years follow-up, 4 years follow-up, 5 years follow-up
  Absence of death from any cause.
Colostomy Free Survival (CFS) | time 0, end of treatment, 6 month post treatment, 1 year follow-up, 2 years follow-up, 3 years follow-up, 4 years follow-up, 5 years follow-up
  Being alive without a temporary or permanent ileostomy or colostomy
Loco-Regional Recurrence (LRR) | time 0, end of treatment, 6 month post treatment, 1 year follow-up, 2 years follow-up, 3 years follow-up, 4 years follow-up, 5 years follow-up
  Presence of disease progression inside the target volume of radiation therapy
Disease-Free Survival (DFS) | time 0, end of treatment, 6 month post treatment, 1 year follow-up, 2 years follow-up, 3 years follow-up, 4 years follow-up, 5 years follow-up
  The time from last treatment to cancer recurrence or death from any cause
Acute toxicity | during treatment, end of treatment
  Acute toxicity caused by chemoradiation according to CTCAE v. 5.0
Late toxicity | 6 month post treatment ,1 year follow-up, 2 years follow-up, 3 years follow-up, 4 years follow-up, 5 years follow-up
  Late toxicity caused by chemoradiation according to CTCAE v. 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Stefania Manfrida, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome, Lazio, Italy